CLINICAL TRIAL: NCT01680445
Title: Observational Telephone Interview Study for Men and Women With Osteoarthritis
Brief Title: Telephone Interview Study for Men and Women With Osteoarthritis
Status: Completed | Type: Observational
Sponsor: Health Outcomes Solutions (Other)
Responsible Party: Principal Investigator, Susan Mathias, Principal Investigator, Health Outcomes Solutions
Other Study IDs: HOS-01-011
Record Dates: First submitted 2011-10-09; First posted 2012-09-07 (Estimated); Last update posted 2012-09-07 (Estimated); Status verified 2012-09

CONDITIONS: Osteoarthritis
Keywords: osteoarthritis, arthritis
MeSH Terms: conditions — Osteoarthritis; Joint Diseases

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The telephone interviews will be conducted to gather information on goal setting and goal attainment from men and women with osteoarthritis.

DETAILED DESCRIPTION:
Interview data used to develop a new self-administered questionnaire

ELIGIBILITY:
Inclusion Criteria:

* Between 40 and 80 years of age
* Have moderate to severe pain
* Diagnosed with osteoarthritis of the hip and/or knee at least 6 months ago
* Currently receiving treatment for osteoarthritis
* Able to speak and read English
* US resident
* Willing to share your thoughts and experiences in a 45-minute telephone interview

Exclusion Criteria:

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: US residents
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2011-03; Primary Completion 2011-04 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Mathias, Principal Investigator — Health Outcomes Solutions
Locations (1):
- Health Outcomes Solutions, Winter Park, Florida, United States